CLINICAL TRIAL: NCT06023303
Title: Prospective Clinical Study to Assess Safety and to Collect Data on Radiofrequency Microneedling Device(s) For the Purpose of Evaluating Treatment on Skin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cynosure, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7043-PM01-2023
Record Dates: First submitted 2023-08-15; First posted 2023-09-05 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Dermatologic Conditions

STUDY DESIGN:
Intervention Model Description: Subjects will be treated with the Potenza device on one side of the face and will receive treatment with Morpheus device on the other side of the face.
Who Masked: Participant
Masking Description: Subjects do not know which side of the face will be treated with either of the devices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A- Split face (Experimental): Group A will receive split face treatments with the Potenza and Morpheus. Randomization will not be used for enrolling subjects to a group but will be used for Group A to determine which side of the face will receive which device.
  Interventions: Device: Potenza; Device: Morpheus
- Group B- none split face (Experimental): Group B will receive treatments on the face, abdomen, and/or back with Potenza and/or Morpheus.
  Interventions: Device: Potenza; Device: Morpheus

INTERVENTIONS:
Device: Potenza — The Radiofrequency microneedling device will be used for treating several skin problems. It is mostly used on the face and neck, specifically to treat jowls and firm the jawline, under aye area, and around the mouth.
Device: Morpheus — The Radiofrequency microneedling device will be used for treating several skin problems. It is mostly used on the face and neck, specifically to treat jowls and firm the jawline, under aye area, and around the mouth.

SUMMARY:
The goal of the Radiofrequency microneedling devices (Potenza and Morpheus) used in this study is to collect clinical data for dermatologic conditions in which electrocoagulation and hemostasis is a viable mechanism for means of improvement.

DETAILED DESCRIPTION:
Up to 20 subjects will be enrolled at 1 study center. Subjects will be enrolled into one of 2 groups. Group A will receive split face treatments with the Potenza and Morpheus. Group B will receive treatments on the face, abdomen, and/or back with Potenza and/or Morpheus. Subjects will attend a screening/pretreatment visit which may be performed on the same day as the treatment visit. Subjects will receive up to 3 treatments with Potenza (and Morpheus).

ELIGIBILITY:
Inclusion Criteria:

* A healthy male or female between the age of 18-65 years old.
* Fitzpatrick skin type I to VI.
* Understands and accepts obligation not to receive any other procedures on the treatment area through the length of the study.
* Understands and accepts the obligation and is logistically able to be present for all visits.
* Is willing to comply with all requirements of the study and sign the informed consent document.

Exclusion Criteria:

* Is pregnant or of childbearing potential and not using medically effective birth control, or has been pregnant in the last 3 months, currently breast feeding or planning a pregnancy during the study.
* The subject is currently enrolled in an investigational drug or device trial or has received an investigational drug or been treated with an investigational device within in the area to be treated 1 month prior to entering this study.
* The subject has received fillers or neurotoxin injections within the past 3 months.
* The subject has a Pacemaker.
* The subject had previous use of gold thread skin rejuvenation.
* The subject has a cut, wound, or infected skin on the area to be treated (but skin eruptions may be treated).
* The subject has a metal implant that interferes with the transmission of energy to the electrical field.
* The subject has any embedded electronic devices that give or receive a signal.
* The subject has Implantable Cardiac Defibrillators (ICD) or Cardiac Resynchronization Therapy (CRT) devices: treatment may interfere with the functionality of the device and/or damage the electronic implant.
* The subject is allergic to adhesives such as glues on medical tape: they should be alerted that a rash may occur on the neutral electronic monitoring pad (NEM or neutral pad) site, and an over-the-counter preparation may be used to treat the area.
* The subject is allergic to gold.
* The subject has an unrealistic expectation of the results: this is not plastic surgery, and all subjects should be fully informed of the treatment's expected results.
* The subject has nerve insensitivity to heat in the treatment area or in the neutral pad placement area.
* The subject has severe laxity or sagging that causes redundant folds of tissue or hanging skin in the area to be treated: this treatment will be ineffective.
* The subject has used Accutane (isotretinoin) six to twelve months prior to treatment, as this can thin the skin and make it brittle.
* The subject is taking aspirin or are currently taking antiplatelets, thrombolytics, anti-inflammatories or anticoagulants.
* The subject has a history of bleeding coagulopathies.
* The subject is allergic to topical anesthetic.
* The subject has keloid formation propensity.
* Subjects with electronic implants such as cardiac defibrillator. It may interfere with the operation of electronic implants or damage the implants, causing risks.
* The subject has any condition or is in a situation which in the investigators opinion may put the subject at significant risk, may confuse study results or may interfere significantly with the subject's participation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-06-21 (Actual); Primary Completion 2023-08-10 (Actual); Study Completion 2023-08-10 (Actual)

PRIMARY OUTCOMES:
Maximum pain reported during treatment. | procedure (during device treatment)
  The maximum pain during treatment per each device will be reported on a scale of 0 (none) to 10 (maximum intolerable pain).

CONTACTS AND LOCATIONS:
Overall Officials: Sean Doherty, Principal Investigator — Cynosure, LLC
Locations (1):
- Cynosure, Inc, Westford, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No